CLINICAL TRIAL: NCT04636047
Title: A Prospective Study on NGS-based Comprehensive Genomic ctDNA Panel in NSCLC Treated With Immunotherapy
Brief Title: NGS-based Comprehensive Genomic ctDNA Panel in NSCLC With Immunotherapy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Lu Shun, Principal Investigator, Shanghai Chest Hospital
Other Study IDs: ShanghaiChest0016
Record Dates: First submitted 2020-09-28; First posted 2020-11-19 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-11

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: The method of gene mutation detection — All samples were detected by NGS CGP panel.

SUMMARY:
Liquid biopsy based on next-generation sequencing (NGS) method has become an increasingly powerful detection tool for clinical research and practice. As a companion diagnostic panel, circulating tumor DNA (ctDNA) assay has the considerable potential to detect the blood tumor mutation burden (bTMB), and bTMB calculated by ctDNA assay is regarded as a novel and promising biomarker for immunotherapy nowadays. Though immune checkpoint inhibitors (ICIs) in immunotherapy are highly effective but can induce severe immune-related adverse events (irAEs), which cannot be better predicted in advance. Meanwhile adoptive transfer of T cells transgenic for tumor-reactive T-cell receptors (TCR) is an attractive immunotherapeutic approach. However, clinical translation is so far limited due to challenges in the identification of suitable target antigens as well as TCRs that are concurrent safe and efficient. Definition of key characteristics relevant for effective and specific tumor rejection is essential to improve current TCR-based immunotherapy. This research is to characterize in-depth TCRs derived from HLA-mismatched allogeneic repertoire targeting different myeloperoxidase (MPO)-derived peptides presented by the same HLA-restriction element. Overall the purpose of this trial is to investigate the combined predictive biomarkers (including bTMB and HLA) related to the immunotherapy effects and the biomarker (TCR) associated with adverse reactions during immunotherapy and hold a predictive role, thus further benefit patients receiving immunotherapy, especially in the advanced stage lung cancer patients where tissue samples are unavailable.

DETAILED DESCRIPTION:
Blood samples including the plasma and PBMC (peripheral blood mononuclear cell) from immunotherapy-naive lung cancer patients will be analyzed by CGP panel (OrigiMed, Inc.) for multiple molecular biomarkers including mutations with sensitivity/resistance to targeted therapies, bTMB, HLA, etc. Treatment methods and outcomes will be followed-up to inspect the clinical benefit and safety with CGP-panel analysis.

ELIGIBILITY:
Inclusion Criteria:

* Participant aged 18 or above, and gender unrestricted
* Individual with pathologically diagnosed lung cancer

Exclusion Criteria:

* Patients with concomitant other tumors
* Individual with severe cardiopulmonary insufficiency and hypoproteinemia
* Women who were pregnant and were during their lactation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients in Shanghai Chest Hospital
Sampling Method: Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2020-11 (Estimated); Primary Completion 2023-02 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | through the whole study period, an average of 3 years
  PFS will be defined as the time from initial treatment to the time of disease progression or death
Blood Tumor Mutational Burden (bTMB) | halfway of the study, an average of 1 year
  bTMB will be defined as the total number of detected somatic mutation counts in coding regions per million bases in plasma ctDNA

SECONDARY OUTCOMES:
Other biomarkers | halfway of the study, an average of 1 year
  The distribution and clinical applications including benefit and adverse reaction of biomarkers such as HLA, TCR and gene mutations in Chinese non-small cell lung cancer patients
Clonality | halfway of the study, an average of 1 year
  The tumor clonality in Chinese non-small cell lung cancer
Overall survival (OS) | through the whole study period, an average of 3 years
  OS will be defined as the time from cancer diagnosed time to the time of death

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China